CLINICAL TRIAL: NCT03739138
Title: A Phase 1/1b, Open-label Clinical Study of Intratumoral/Intralesional Administration of MK-4621/JetPEI as Monotherapy or in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic or Recurrent Solid Tumors
Brief Title: Intratumoral/Intralesional Administration of MK-4621/JetPEI™ With or Without Pembrolizumab in Participants With Advanced/Metastatic or Recurrent Solid Tumors (MK-4621-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4621-002; MK-4621-002 (Other: Merck Protocol Number); 2018-000845-37 (EudraCT Number)
Record Dates: First submitted 2018-07-31; First posted 2018-11-13 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumors
Keywords: Programmed Death-1 (PD-1, PD1),; Programmed Death-Ligand 1 (PD-L1, PDL1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MK-4621 Monotherapy (Arm 1) (Experimental): Participants receive MK-4621 once a week (Q1W) during each 21-day cycle for a maximum duration of 6 cycles.
  Interventions: Biological: MK-4621
- MK-4621 + Pembrolizumab (Arm 2) (Experimental): Participants receive escalating doses of MK-4621 Q1W during each 21-day cycle for a maximum duration of 6 cycles in combination with pembrolizumab at a fixed dose 200 mg every 3 weeks (Q3W) for a maximum duration of 6 cycles. Participants may continue on treatment with pembrolizumab after Cycle 6 for up to 35 cycles (Cycles 7-35, approximately 2 years) from the start of treatment. Dose escalation of MK-4621 will be based on safety and tolerability.
  Interventions: Biological: MK-4621; Biological: Pembrolizumab
- Intrahepatic MK-4621 + Pembrolizumab (Arm 3) (Experimental): Participants receive MK-4621 as monotherapy on Day 1 only of the first 21-day cycle (run-in phase). After the run-in phase, participants receive escalating doses of MK-4621 Q3W in combination with pembrolizumab at a fixed dose 200 mg Q3W for a maximum duration of 5 cycles (Cycles 2-6). Participants may continue on treatment with pembrolizumab for up to 35 cycles (Cycles 7-35, approximately 2 years) from the start of treatment. Dose escalation of MK-4621 will be based on safety and tolerability.
  Interventions: Biological: MK-4621; Biological: Pembrolizumab

INTERVENTIONS:
Biological: MK-4621 — MK-4621 is delivered via the JetPEI™ in vivo linear polyethylenimine nucleic acid delivery system as follows:
  For Arm 1: administered intratumorally Q1W, on Days 1, 8, and 15 of each 21-day cycle.
  For Arm 2: administered intratumorally Q1W, on Days 1, 8, and 15 of each 21-day cycle according to randomization.
  For Arm 3: administered intratumorally Q3W, on Day 1 of each 21-day cycle. Range administered will depend upon allocation and be based on emerging safety data.
Biological: Pembrolizumab — 200 mg administered intravenously (IV) on Day 1 of each 21-day cycle beginning with Cycle 1 (Arm 2) or Cycle 2 (Arm 3).
  Arms: Intrahepatic MK-4621 + Pembrolizumab (Arm 3); MK-4621 + Pembrolizumab (Arm 2)

SUMMARY:
The purpose of this study is to evaluate safety and tolerability, pharmacokinetics (PK), and preliminary antitumor activity of intratumoral (IT) / intralesional injections of MK-4621 delivered via the JetPEI™ in vivo linear polyethylenimine nucleic acid delivery system as monotherapy and in combination with pembrolizumab in participants with advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically- or cytologically-confirmed advanced/metastatic solid tumor by pathology report and has received, or been intolerant to, all treatment known to confer clinical benefit
* Has submitted an evaluable baseline tumor sample for analysis before start of treatment
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Demonstrates adequate organ function
* Male participants must agree to use approved contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period
* Female participants who are not pregnant or breastfeeding, and who are either not a woman of childbearing potential (WOCBP), or are a WOCBP who agrees to use approved contraception during the treatment period and for at least 120 days after the last dose of study treatment

Arms 1 and 2: have 3 lesions defined as follows: 1) at least 1 cutaneous or subcutaneous lesion that is amenable to injection and biopsy (lesion 1) that is measurable as defined by RECIST 1.1, 2) at least 1 discrete non-injected, non-biopsied lesion that is measurable as defined by RECIST 1.1 (lesion 2), and 3) at least 1 discrete and/or distant non-injected lesion amenable for biopsy (lesion 3)

Arm 3 only: Has metastatic liver and/or liver lesion involvement that does not exceed one third of the total liver volume in participants to be treated by liver IT injection. Hepatocellular carcinoma participants are excluded from eligibility of intratumoral liver injection. For Arm 3, at least 2 lesions have to be identified as follows: 1) at least 1 liver lesion amenable to image-guided intratumoral injection and biopsy via ultrasound guidance or cross-sectional imaging (CT/MRI) guidance and must be measurable as defined by RECIST 1.1 (lesion 1) and 2) at least 1 other discrete non-injected, non-biopsied lesion that is measurable as defined by RECIST 1.1 (lesion 2)

Exclusion Criteria:

* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks prior to the first dose of study therapy, or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from any AEs that were due to cancer therapeutics administered more than 4 weeks earlier
* History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* Has hepatocellular carcinoma (for Arm 3 only)
* Has clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has had a severe hypersensitivity reaction to treatment with a monoclonal antibody/components of the study treatment
* Has an active infection requiring therapy
* Has history of interstitial lung disease
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a known history of human immunodeficiency virus (HIV) infection and/or Hepatitis B or C infections, or known to be positive for Hepatitis B surface antigen (HBsAg)/Hepatitis B virus (HBV) DNA or Hepatitis C Antibody or RNA
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorder that would interfere with cooperating with the requirements of the study
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Has not fully recovered from any effects of major surgery without significant detectable infection
* WOCBP who has a positive urine pregnancy test within 72 hours before the first dose of study treatment
* Has received a live-virus vaccine within 30 days of planned treatment start
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Prior exposure to immunotherapeutics is allowed, including PD-1 and PD-L1 inhibitors, provided participant did not experience a ≥Grade 3 drug-related toxicity on monotherapy with a PD-1 or PD-L1 inhibitor
* Has a history of re-irradiation for squamous cell carcinoma of head and neck (SCCHN) at the projected injection site
* Has a tumor(s) in direct contact or encases a major blood vessel and has ulceration and/or fungation onto the skin surface

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (9):
- France (4):
  - Institut Bergonie ( Site 3303), Bordeaux
  - CHU La Timone ( Site 3304), Marseille
  - Institut Curie ( Site 3302), Paris
  - Institut Gustave Roussy ( Site 3301), Villejuif
- Germany (2):
  - Charite Campus Benjamin Franklin ( Site 4903), Berlin
  - Universitaetsklinikum Carl Gustav Carus der TU Dresden ( Site 4901), Dresden
- Spain (2):
  - Hospital Universitario Fundacion Jimenez Diaz ( Site 3401), Madrid
  - Centro Integral Oncologico Clara Campal START Madrid ( Site 3402), Madrid
- Oxford University Hospital NHS Foundation Trust ( Site 4401), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Moreno V, Calvo E, Middleton MR, Barlesi F, Gaudy-Marqueste C, Italiano A, Romano E, Marabelle A, Chartash E, Dobrenkov K, Zhou H, Connors EC, Zhang Y, Wermke M. Treatment with a retinoic acid-inducible gene I (RIG-I) agonist as monotherapy and in combination with pembrolizumab in patients with advanced solid tumors: results from two phase 1 studies. Cancer Immunol Immunother. 2022 Dec;71(12):2985-2998. doi: 10.1007/s00262-022-03191-8. Epub 2022 May 21. PMID 35596791

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 30 participants were enrolled to Arm 2 at 3 different dose levels. The study was terminated before enrolment into Arm 1 and Arm 3.
Groups:
- MK-4621 Monotherapy (Arm 1): Participants were to receive MK-4621 monotherapy once a week (Q1W) during each 21-day cycle for a maximum duration of 6 cycles. No participants were enrolled in this arm.
- MK-4621 0.4 mg + Pembrolizumab (Arm 2): Participants received MK-4621 0.4 mg Q1W during each 21-day cycle for a maximum duration of 6 cycles in combination with pembrolizumab at a fixed dose 200 mg every 3 weeks (Q3W) for a maximum duration of 6 cycles. Participants could continue to receive pembrolizumab monotherapy after Cycle 6 for up to 35 cycles (Cycles 7-35, approximately 2 years) from the start of treatment.
- MK-4621 0.6 mg + Pembrolizumab (Arm 2): Participants received MK-4621 0.6 mg Q1W during each 21-day cycle for a maximum duration of 6 cycles in combination with pembrolizumab 200 mg Q3W for a maximum duration of 6 cycles. Participants could continue to receive pembrolizumab monotherapy after Cycle 6 for up to 35 cycles (Cycles 7-35, approximately 2 years) from the start of treatment.
- MK-4621 0.8 mg + Pembrolizumab (Arm 2): Participants received MK-4621 0.8 mg Q1W during each 21-day cycle for a maximum duration of 6 cycles in combination with pembrolizumab 200 mg Q3W for a maximum duration of 6 cycles. Participants could continue to receive pembrolizumab monotherapy after Cycle 6 for up to 35 cycles (Cycles 7-35, approximately 2 years) from the start of treatment.
- Intrahepatic MK-4621 + Pembrolizumab (Arm 3): Participants were to receive MK-4621 monotherapy via intrahepatic administration on Day 1 only of the first 21-day cycle (run-in phase). After the run-in phase, participants were to receive MK-4621 Q3W in combination with pembrolizumab 200 mg Q3W for a maximum duration of 5 cycles (Cycles 2-6). No participants were enrolled in this arm.
Period: Overall Study
Arm/Group | MK-4621 Monotherapy (Arm 1) | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2) | Intrahepatic MK-4621 + Pembrolizumab (Arm 3)
Started | 0 | 7 | 5 | 18 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 7 | 5 | 18 | 0
Not completed — Death | 0 | 7 | 4 | 13 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2) | Total
Number analyzed (Participants) | 7 | 5 | 18 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (10.1) | 61.2 (13.8) | 57.7 (10.5) | 58.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 8 | 18
  Male | 1 | 1 | 10 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 10 | 18
  Unknown or Not Reported | 1 | 3 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 3 | 13 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: The following toxicities during DLT evaluation period were considered DLT, if assessed by investigator to be possibly, probably, or definitely related to treatment: Grade (Gr) 4 nonhematologic toxicity; Gr 4 hematologic toxicity lasting ≥7 days or protocol-specified thrombocytopenia; any nonhematologic adverse event (AE) ≥Gr 3 in severity (with exceptions); any Gr 3/Gr 4 nonhematologic laboratory value if clinically significant medical intervention was required to treat the participant, or the abnormality led to hospitalization, or the abnormality persisted for >1 week; or the abnormality resulted in a drug-induced liver injury; febrile neutropenia Gr 3/Gr 4; >2 week delay in initiating Cycle 2 due to treatment-related toxicity; any treatment-related toxicity that caused the participant to discontinue treatment during Cycle 1; missing >2 injections of MK-4621 during Cycle 1, or Gr 5 toxicity. The percentage of participants who experienced DLTs were reported for each arm.
Time Frame: Up to 21 days (Cycle 1)
Population: The DLT-evaluable population included all randomized participants who received at least 1 dose of study treatment and who met the criteria for DLT evaluability (e.g. completed the DLT evaluation period without a DLT or experienced a DLT in the DLT evaluation period).
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2)
Number analyzed (Participants) | 7 | 5 | 18
Percentage of Participants | 0.0 [0.0 to 18.2] | 0.0 [0.0 to 23.5] | 5.6 [1.1 to 15.5]

2. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant that was temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experienced an AE was reported for each arm.
Time Frame: Up to approximately 13 months
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2)
Number analyzed (Participants) | 7 | 5 | 18
Participants | 7 | 5 | 18

3. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant that was temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who discontinued study treatment due to an AE was reported for each arm.
Time Frame: Up to approximately 13 months
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2)
Number analyzed (Participants) | 7 | 5 | 18
Participants | 0 | 0 | 2

4. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of MK-4621
Description: AUC is the area under the plot of plasma concentration of drug against time after drug administration and is of particular use in estimating bioavailability of drugs, and in estimating total clearance of drugs. Blood samples were collected at multiple time points (pre-dose and post-dose) during the study to assess the AUC of MK-4621.
Time Frame: Day 1 of 21-day Cycles 1 and 2: pre-dose (1-8 hours), end of IT injection up to +5 minutes (0.0 hours), 0.5, 1.0, 2, 4, and 6 hours. Samples also collected at 24 hours after MK-4621 dose for Cycle 1 Day 1 only.
Population: The Per Protocol population included all randomized participants who received at least 1 dose of study treatment, who complied with the protocol with no protocol deviations, and who had available data for pharmacokinetic measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2)
Number analyzed (Participants) | 7 | 5 | 18
h*ng/mL | NA (NA) — NA = Noncompartmental AUC could not be calculated due to MK-4621 plasma concentrations that were below level of quantitation (BLOQ) for most participants. | NA (NA) — NA = Noncompartmental AUC could not be calculated due to MK-4621 plasma concentrations that were BLOQ for most participants. | NA (NA) — NA = Noncompartmental AUC could not be calculated due to MK-4621 plasma concentrations that were BLOQ for most participants.

5. Secondary Outcome: Minimum Concentration (Cmin) of MK-4621
Description: Cmin was defined as the minimum or "trough" concentration of MK-4621 observed after its administration and just prior to the administration of a subsequent dose. Blood samples were collected at multiple time points (pre-dose and post-dose) during the study to assess the Cmin of MK-4621.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2)
Number analyzed (Participants) | 7 | 5 | 18
ng/mL | NA (NA) — NA = Noncompartmental Cmin could not be calculated due to MK-4621 plasma concentrations that were BLOQ for most participants. | NA (NA) — NA = Noncompartmental Cmin could not be calculated due to MK-4621 plasma concentrations that were BLOQ for most participants. | NA (NA) — NA = Noncompartmental Cmin could not be calculated due to MK-4621 plasma concentrations that were BLOQ for most participants.

6. Secondary Outcome: Maximum Concentration (Cmax) of MK-4621
Description: Cmax was defined as the maximum or "peak" concentration of MK-4621 observed after its administration. Blood samples were collected at multiple time points (pre-dose and post-dose) to assess the Cmax of MK-4621.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2)
Number analyzed (Participants) | 7 | 5 | 18
ng/mL | NA (NA) — NA = Noncompartmental Cmax could not be calculated due to MK-4621 plasma concentrations that were BLOQ for most participants. | NA (NA) — NA = Noncompartmental Cmax could not be calculated due to MK-4621 plasma concentrations that were BLOQ for most participants. | NA (NA) — NA = Noncompartmental Cmax could not be calculated due to MK-4621 plasma concentrations that were BLOQ for most participants.

7. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR, disappearance of all evidence of disease) or Partial Response (PR, ≥30% decrease in the sum of diameters of target lesions) as assessed by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) based upon investigator assessment. ORR was reported for each treatment arm.
Time Frame: Up to approximately 22 months (through data cut-off of 02-Mar-2021)
Population: All randomized participants who received at least 1 dose of study treatment and had a baseline scan that demonstrated measurable disease by the investigator's assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2)
Number analyzed (Participants) | 7 | 5 | 18
Percentage of Participants | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 52.2] | 16.7 [3.6 to 41.4]

ADVERSE EVENTS:
Time Frame: Up to approximately 22 months (through data cut-off of 02-Mar-2021)
Description: All-Cause Mortality table includes all randomized participants. Serious and Other AE tables include all randomized participants who received at least 1 dose of study drug. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" unrelated to drug were excluded as AEs.
Arm/Group | MK-4621 0.4 mg + Pembrolizumab (Arm 2) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) | MK-4621 0.8 mg + Pembrolizumab (Arm 2)
All-Cause Mortality (participants affected / at risk) | 7/7 | 4/5 | 13/18
Serious Adverse Events (participants affected / at risk) | 6/7 | 3/5 | 11/18
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-4621 0.4 mg + Pembrolizumab (Arm 2) (N=7) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) (N=5) | MK-4621 0.8 mg + Pembrolizumab (Arm 2) (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (2) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-4621 0.4 mg + Pembrolizumab (Arm 2) (N=7) | MK-4621 0.6 mg + Pembrolizumab (Arm 2) (N=5) | MK-4621 0.8 mg + Pembrolizumab (Arm 2) (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 6 (7)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (6)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dental paraesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 2 (2) | 4 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5)
Asthenia (General disorders) | 0 (0) | 1 (1) | 3 (5)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 3 (4) | 2 (4) | 6 (10)
Extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (4) | 1 (1) | 4 (4)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 2 (6)
Implant site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 4 (5)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 4 (5) | 10 (39)
Cytokine release syndrome (Immune system disorders) | 1 (2) | 0 (0) | 4 (19)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injection site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (4)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Tri-iodothyronine free decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (5) | 0 (0) | 2 (3)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT03739138/Prot_SAP_000.pdf